CLINICAL TRIAL: NCT05006742
Title: Comparison of Transbronchial Cryobiopsy and Forceps Biopsy in Lung Transplant Recipients: A Prospective Analysis for Acute Cellular Rejection
Brief Title: Comparison of Transbronchial Cryobiopsy and Forceps Biopsy in Lung Transplant Recipients
Acronym: Kryo-LUTPL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Carolin Steinack, principal investigator, University of Zurich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ID 2021-00466
Record Dates: First submitted 2021-07-31; First posted 2021-08-16 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Lung Transplant Rejection; Lung Transplant Failure and Rejection
Keywords: Cryobiopsy; Transbronchial Biopsy
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Intervention Model Description: This is a prospective randomized trial to assess diagnostic accuracy and safety of cryobiopsy using two different transbronchial biopsy techniques. Included patients are 1:1 randomized to receive either cryobiopsy (CB study arm) or forceps biopsy and cryobiopsy within the same session (FB-CB study arm). Both, forceps biopsy and cryobiopsy are performed according to official recommendations. The biopsies will be scored for ACR according to the ISHLT criteria (A0 - A4) by 3 pathologists. A subgroup analysis in the FB-CB study arm will compare FB and CB of the same patient in order to prevent second bronchoscopy due to inconclusive histological result of FB and lung function decline being suspicious for ACR.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CB study arm (Active Comparator): Included patients are 1:1 randomized to receive either CB (CB study arm) or FB and CB within the same session (FB-CB study arm
  Interventions: Procedure: CB study arm
- FB-CB study arm (Active Comparator): Included patients are 1:1 randomized to receive either CB (CB study arm) or FB and CB within the same session (FB-CB study arm
  Interventions: Procedure: FB-CB study arm

INTERVENTIONS:
Procedure: CB study arm — Included patients are randomized to receive cryobiopsy
  Arms: CB study arm
Procedure: FB-CB study arm — Included patients are randomized to receive forceps biopsy and cryobiopsy within the same session
  Arms: FB-CB study arm

SUMMARY:
CLAD is defined as loss of lung function after other factors, particularly infections have been excluded. Readily accessible diagnostic procedures to detect acute cellular rejection at the earliest possible occasion is crucial for posttransplant survival. Serial lung function tests, laboratory testing and pulmonary imaging are only clinical indicators of chronic allograft dysfunction in lung transplant recipients. Since forceps biopsy to detect acute cellular rejection in lung transplant recipients has several shortcomings, the purpose of this study is to investigate a new biopsy technique using the transbronchial cryoprobe.

DETAILED DESCRIPTION:
Eventually, histopathological confirmation is indispensable to establish the diagnosis of acute cellular rejection. The current gold standard for diagnosis and grading of acute cellular rejection in order to initialize the optimal treatment, with particular regard to adjusting immunosuppression, is forceps biopsy to obtain ≥ five samples. Forceps biopsy has a reasonable risk profile in experienced centers and is performed 2, 4, 6 and 12 months posttransplant and when indicated. Given these concerns about diagnostic yield in forceps biopsy and unjustifiable risks after surgical lung biopsy, cryobiopsy has arisen as promising alternative diagnostic procedure. The value of cryobiopsy to obtain a conclusive diagnosis of ACR is discussed controversially due the lack of safety and efficacy data in lung transplant recipients

ELIGIBILITY:
Inclusion Criteria:

* routinely performed surveillance bronchoscopy and when indicated including serial FB and CB in the same session in patients wo had undergone lung transplant
* male or female subject of at least 18 years of age
* written informed consent after participant's information signed by patient

Exclusion Criteria:

* age < 18 years
* Lacking ability to form an informed consent (including impaired judgement, communication barriers)
* Contraindication against bronchoscopy (e.g. co-morbidities)
* INR > 2 or Thrombocytes < 50000
* Double antiplatelet drugs (e.g. ASS and Clopidogrel) within 7 days before biopsy
* Anticoagulation with NOAK within 48 hours before biopsy
* Moderate or severe pulmonary hypertension (mPAP > 30 mmHg, RV/RA >30 mmHg)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
diagnostic yield | up to 1 month
  To investigate the diagnostic yield of two different transbronchial lung biopsy techniques (forceps and cryobiopsy) for diagnosis of acute cellular rejection in lung transplant recipients.

SECONDARY OUTCOMES:
% of patients with treatment alteration due to the biopsy result | up to 1 month
  Impact on treatment decisions depending of the pathology results
Incidence of treatment-emergent adverse events as assessed by pneumothorax rate | up to 1 week
  data on safety
Incidence of treatment-emergent adverse events as assessed by bleeding events | up to 1 week
  data on safety
interobserver agreement between 3 pathologists | up to 3 months
  The biopsies are assessed for acute cellular rejection by three pathologists.

CONTACTS AND LOCATIONS:
Overall Officials: Carolin Steinack, Principal Investigator — University of Zurich
Locations (1):
- University hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yarmus L, Akulian J, Gilbert C, Illei P, Shah P, Merlo C, Orens J, Feller-Kopman D. Cryoprobe transbronchial lung biopsy in patients after lung transplantation: a pilot safety study. Chest. 2013 Mar;143(3):621-626. doi: 10.1378/chest.12-2290. PMID 23328889
- [Result] Fruchter O, Fridel L, Rosengarten D, Raviv Y, Rosanov V, Kramer MR. Transbronchial cryo-biopsy in lung transplantation patients: first report. Respirology. 2013 May;18(4):669-73. doi: 10.1111/resp.12037. PMID 23294256
- [Result] Roden AC, Kern RM, Aubry MC, Jenkins SM, Yi ES, Scott JP, Maldonado F. Transbronchial Cryobiopsies in the Evaluation of Lung Allografts: Do the Benefits Outweigh the Risks? Arch Pathol Lab Med. 2016 Apr;140(4):303-11. doi: 10.5858/arpa.2015-0294-OA. Epub 2015 Oct 21. PMID 26488148
- [Result] Gershman E, Ridman E, Fridel L, Shtraichman O, Pertzov B, Rosengarten D, Rahman NA, Shitenberg D, Kramer MR. Efficacy and safety of trans-bronchial cryo in comparison with forceps biopsy in lung allograft recipients: Analysis of 402 procedures. Clin Transplant. 2018 Apr;32(4):e13221. doi: 10.1111/ctr.13221. Epub 2018 Feb 28. PMID 29436115